CLINICAL TRIAL: NCT03049943
Title: Different Low Level Laser Protocols for Therapy of Hyposalivation
Brief Title: Low Level Laser Therapy for Hyposalivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Assisstant Professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/05/2012
Record Dates: First submitted 2017-02-03; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Hyposalivation
Keywords: low level laser therapy; hyposalivation
MeSH Terms: conditions — Xerostomia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser wavelength of 830 nm (Active Comparator): This group comprised 15 female patients with hyposalivation whose major salivary glands were treated for 10 consecutive days with low level laser therapy of 830 nm.The whole unstimulated and stimulated saliva was measured each day during 10 days, before and after laser treatment and 10th day after treatment was ended.
  Interventions: Device: low level laser
- Laser wavelength of 685 nm (Experimental): This group comprised 15 female patients with hyposalivation whose major salivary glands were treated for 10 consecutive days with low level laser therapy of 685 nm.The whole unstimulated and stimulated saliva was measured each day during 10 days, before and after laser treatment and 10th day after treatment was ended.
  Interventions: Device: low level laser

INTERVENTIONS:
Device: low level laser

SUMMARY:
The aim of this study was to compare the effects of different wave lengths of LLLT on salivation in participants suffering from hyposalivation.

This study included 30 participants whose major salivary glands were treated with low intensity diode laser BTL2000 (Medical Technologies, s.r.o., Czech Republic) during 10 consecutive days. Patients were randomly assigned in two groups, each of 15 patients, and treated with LLLT of 830 nm and LLLT of 685 nm, respectively. The whole unstimulated and stimulated saliva was measured each day during 10 days, before and after laser treatment and 10th day after treatment was ended.

DETAILED DESCRIPTION:
Low level laser treatment has proved to be effective for a wide range of oral pathologies including oral dryness, but the literature still lacks reports of clinical trials and protocols. The aim of this study was to evaluate the effects of two different laser wave lengths on salivation of patients suffering from hyposalivation. This with purpose to possibly find the optimum laser wavelength for the treatment, and to determine the better protocol for the patients suffering from hyposalivation. This study included 30 patients whose major salivary glands were treated with low intensity diode laser BTL2000 (Medical Technologies, s.r.o., Czech Republic) during 10 consecutive days. Patients were randomly assigned in two groups, each of 15 patients, and treated with LLLT of 830 nm and LLLT of 685 nm, respectively. The whole unstimulated and stimulated saliva was measured in graduated tubes each day during 10 days, before and after laser treatment and 10th day after treatment was ended.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from hyposalivation, with medical histories free of radiotherapy and Sjögren's syndrome

Exclusion Criteria:

* medical histories of radiotherapy and Sjögren's syndrome

Ages: 52 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2014-09-16 (Actual); Study Completion 2014-09-16 (Actual)

PRIMARY OUTCOMES:
Difference in average salivary flow rate, before and after low level laser treatment | 10 days
  The whole unstimulated and stimulated saliva was measured each day during 10 days, before and after laser treatment

SECONDARY OUTCOMES:
Average salivary flow rate | 1 day (Average salivary flow rate 10th day after the end of LLLT)
  Average salivary flow rate 10th day after the end of LLLT

CONTACTS AND LOCATIONS:
Overall Officials: Božana Lončar Brzak, Assist.Prof., Principal Investigator — School of Dental Medicine, University of Zagreb
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Loncar B, Stipetic MM, Baricevic M, Risovic D. The effect of low-level laser therapy on salivary glands in patients with xerostomia. Photomed Laser Surg. 2011 Mar;29(3):171-5. doi: 10.1089/pho.2010.2792. Epub 2010 Nov 6. PMID 21054200